CLINICAL TRIAL: NCT04090632
Title: Impact of Anthropometrics Data and of Physical Activity Level in Closed kineTic Chain Upper Extremity Stability Test (CKCUEST) - EPOLTEST Study
Brief Title: Impact of Anthropometrics Data and of Physical Activity Level in Closed kineTic Chain Upper Extremity Stability Test
Acronym: EPOLTEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC19.0147
Record Dates: First submitted 2019-08-12; First posted 2019-09-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2020-06

CONDITIONS: Shoulder Pain
Keywords: CKCUEST; Physical activity; rehabilitation
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a monocentric interventional prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- closed kineTic chain upper Extremity Stability Test (Experimental): Each patient receive the same intervention, the CKCUEST. The CKCUEST is a functional test which assess shoulder's stability. Patient is in push-up position, with 91 cm between his hands. His body is straight and his foots are squeeze. patient has to touch his hand with his other one and returns in the initial position. Then, patient repeats this movement with his other hand, etc, during 15 secondes. The CKCUEST score is the movement's number performed.
  Interventions: Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test

INTERVENTIONS:
Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test — Each patient receive the same intervention, the CKCUEST. The CKCUEST is a functional test which assess shoulder's stability. Patient is in push-up position, with 91 cm between his hands. His body is straight and his foots are squeeze. patient has to touch his hand with his other one and returns in the initial position. Then, patient repeats this movement with his other hand, etc, during 15 secondes. The CKCUEST score is the movement's number performed.

SUMMARY:
The purpose of this study is to evaluate impact of anthropometric criteria to CKCUEST score.

ELIGIBILITY:
Inclusion Criteria:

* Aged to 18 to 25 years
* Capacity to consent
* Who has signed the consent

Exclusion Criteria:

* fracture history or upper limb luxation
* is not possible to do the test because of pain
* pregnant or nursing
* refuse to participate
* guardianship or protection of vulnerable adult

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) score | Day 1
  Closed Kinetic Chain Upper Extremity Stability Test/ The CKCUEST is a functional test which assess shoulder's stability. Patient is in push-up position, with 91 cm between his hands. His body is straight and his foots are squeeze. patient has to touch his hand with his other one and returns in the initial position. Then, patient repeats this movement with his other hand, etc, during 15 secondes. The CKCUEST score is the movement's number performed. The outcome measure will be the mean of the three test realisation.

SECONDARY OUTCOMES:
Global Physical Activity Questionnaire (GPAQ) | Day 1
  Global Physical Activity Questionnaire. It is a standardized questionnaire which evaluate the global physical activity. GPAQ takes into account both number and intensity of activity. There are 4 parts (profession activities,day to day ways of moving, hobbies, sedentarity) in total being 16 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, Finistère, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Result] Lepinet U, Tanniou J, Communier EC, Creach V, Beaumont M. Impact of anthropometric data and physical activity level on the closed kinetic chain upper extremity stability test (CKCUEST) score: A cross-sectional study. Phys Ther Sport. 2023 Nov;64:91-96. doi: 10.1016/j.ptsp.2023.09.004. Epub 2023 Sep 27. PMID 37806101